CLINICAL TRIAL: NCT02659826
Title: Effects of Non-invasive Stimulation on Central Nervous System Excitability of Healthy Volunteers
Brief Title: Non-invasive Stimulation on Central Nervous System Excitability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, PhD, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NIS_CNSexcitability
Record Dates: First submitted 2015-10-19; First posted 2016-01-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: Transcutaneous spinal direct current stimulation; Transcranial Magnetic Stimulation; Gait Training; Central Nervous System Excitability; Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- anodal tsDCS and gait training (Experimental): Volunteers will be submitted to anodal transcutaneous spinal cord stimulation and gait training
  Interventions: Device: anodal tsDCS; Device: Gait training
- cathodal tsDCS and gait training (Experimental): Volunteers will be submitted to cathodal transcutaneous spinal cord stimulation and gait training
  Interventions: Device: cathodal tsDCS; Device: Gait training
- sham tsDCS and gait training (Sham Comparator): Volunteers will be submitted to sham transcutaneous spinal cord stimulation and gait training
  Interventions: Device: sham tsDCS; Device: Gait training
- High frequency rTMS and gait training (Experimental): Volunteers will be submitted to high frequency transcranial magnetic stimulation and gait training
  Interventions: Device: Gait training; Device: High frequency rTMS
- Low frequency rTMS and gait training (Experimental): Volunteers will be submitted to low frequency transcranial magnetic stimulation and gait training
  Interventions: Device: Gait training; Device: Low frequency rTMS
- sham rTMS and gait training (Sham Comparator): Volunteers will be submitted to sham transcranial magnetic stimulation and gait training
  Interventions: Device: Gait training; Device: sham rTMS

INTERVENTIONS:
Device: anodal tsDCS — Transcutaneous spinal cord stimulation will be delivered through a direct current (DC) stimulator (NeuroConn Plus, Germany) using a pair of saline-soaked sponge electrodes (35cm²). The active electrode (anode) will be placed between the eleventh and the twelfth thoracic vertebra) and the reference electrode, over the right arm (deltoid muscle). Will be delivered a current intensity of 2.5 milliampere (mA), fade in and fade out of 10 seconds, during 20 minutes.
  Arms: anodal tsDCS and gait training
Device: cathodal tsDCS — Transcutaneous spinal cord stimulation will be delivered through a DC stimulator (NeuroConn Plus, Germany) using a pair of saline-soaked sponge electrodes (35cm²). The active electrode (cathode) will be placed between the eleventh and the twelfth thoracic vertebra) and the reference electrode, over the right arm (deltoid muscle). Will be delivered a current intensity of 2.5 mA, fade in and fade out of 10 seconds, during 20 minutes.
  Arms: cathodal tsDCS and gait training
Device: sham tsDCS — sham transcutaneous spinal cord stimulation will be delivered through a DC stimulator (NeuroConn Plus, Germany) using a pair of saline-soaked sponge electrodes (35cm²). The electrode anode will be placed between the eleventh and the twelfth thoracic vertebra) and the reference electrode, over the right arm (deltoid muscle). Will be delivered a current intensity of 2.5 mA, fade in and fade out of 10 seconds, during only 30 seconds but the volunteers will continue with electrodes montage for 20 minutes.Thus, early sensations (eg. mild to moderate tingling or itch) on stimulation site will be experienced without inducing any modulatory effects.
  Arms: sham tsDCS and gait training
Device: Gait training — It consists of moderate gait training exercise for 20 minutes. To ensure that the exercise will be performed at moderate intensity will be used the 64% - 76% of maximum heart rate (HRmax = 220-age). Heart rate will be monitored every three minutes through a heart polar. In addition will be monitored perceived effort, gait speed and inclination of the treadmill. The Borg scale will be used to evaluate perceived effort. This is an analogue scale graded from 6 (light exercise) to 20 points (exhaustive exercise). Information about the exercise on the treadmill will be noted in the evolution record.
Device: High frequency rTMS — Initially, the higher cortical representation area (hotspot) of first right dorsal interosseous (FDI) muscle will be determined through a figure-eight coil connected to the magnetic stimulator (Rapid2, Magstim, UK) held manually and positioned over the scalp (C3 - 10/20 System) at an angle of 45 degrees from the midline pointed to the target muscle (FDI). Thereafter, RMT will be measure. rTMS protocols was based on previous studies. High frequency protocol: 20 hertz (Hz), 90% RMT, 45 trains, 40 stimuli per train, inter interval of 28 seconds, 1800 stimuli. After each rTMS session, presence of adverse effects will be computed.
  Arms: High frequency rTMS and gait training
Device: Low frequency rTMS — Initially, the higher cortical representation area (hotspot) of first right dorsal interosseous (FDI) muscle will be determined through a figure-eight coil connected to the magnetic stimulator (Rapid2, Magstim, UK) held manually and positioned over the scalp (C3 - 10/20 System) at an angle of 45 degrees from the midline pointed to the target muscle (FDI). Thereafter, RMT will be measure. Low frequency protocol: 1Hz, 90% RMT, 1500 stimuli (1 train). After each rTMS session, presence of adverse effects will be computed.
  Arms: Low frequency rTMS and gait training
Device: sham rTMS — The hotspot of first right dorsal interosseous (FDI) muscle will be determinate through a figure-eight coil connected to the magnetic stimulator positioned over the motor primary cortex (C3). Then, the motor threshold (RMT) of FDI will be measure. Sham rTMS will be performed with low frequency (1Hz, 90% RMT, 1500 stimuli) protocol using two coils. The first one - connected to the stimulator - will be positioned on a coil support close to the volunteer but not visible. Therefore, characteristic stimulation noises will be audible. The second - disconnected to the stimulator - will be placed over left primary motor area. After each rTMS session, presence of adverse effects will be computed.
  Arms: sham rTMS and gait training

SUMMARY:
A crossover trial with healthy volunteers will be conducted. Six sessions will be performed once a week in a counterbalanced order and at least with seven days washout period to minimize carry-over effects. In each session, volunteers will be submitted to quantity and quality of sleep, type of eating, fatigue and motivation level, cortical brain activity measures through paired pulse transcranial magnetic stimulation (ppTMS), spinal cord activity measures through electrical stimulation, non-invasive spinal stimulation (tsDCS) or non-invasive brain stimulation (rTMS) and physical exercise (gait training).

DETAILED DESCRIPTION:
After given prior informed consent, volunteers will be submitted to six pseudorandomized sessions using a website (randomization.com) by a non-involved researcher. At study beginning, volunteers will be evaluated through structured questionnaire and each session, will comprise the following experimental sequence:

1. Quantity and quality of sleep: It will be enquired how many hours the volunteer slept in the last night. The quality of the sleep will be measured through an analogue scale graded from 0 (worst quality of sleep) to 10 points (best quality of sleep).
2. Type of eating: All the individuals will be asked about ingestion of food and drinks that could change the cortical excitability ( e. g.; coffee, chocolate, energetic, soda e etcc). If positive, researchers will record the time since of ingestion and quantify the amount of food.
3. Fatigue and motivation level: Fatigue and motivation level: Fatigue and motivation levels: It will be measured through an analogue scale graded from 0 (lower fatigue or motivation levels) to 10 points (greater fatigue or motivation levels).
4. Cortical excitability: the cortical will be measured through the motor evoked potential (MEP), short intracortical inhibition (SICI) and intracortical facilitation (ICF). All the measures will be evaluated through transcranial magnetic stimulation (Neurosoft, Russia). Initially, rest motor threshold (RMT) will be determined by finding the lowest stimulator output that elicit motor evoked potential (MEP) at least 50 microvolts (μV). For RMT measure, a figure-eight coil connected to the magnetic stimulator held manually at 45 degrees from the midline, will be placed over the right primary motor cortex (C3 - 10/20 System). The short intracortical inhibition (SICI) and intracortical facilitation (ICF) will be evaluated by paired pulse transcranial magnetic stimulation. A subthreshold conditioning stimuli (80% of RMT) and suprathreshold test stimuli (130% of RMT) will be delivered at an interstimulus interval (ISI) of 2 milliseconds for SICI and 10 milliseconds for ICF. Ten stimuli will be applied at each condition (unconditioned pulse and pairs of stimuli with ISI of 3 and 20 milliseconds). Stimuli order delivery will be pseudo-randomized and SICI and ICF will be expressed as conditioned stimulus percentage regarding unconditioned stimulus. The MEP value will be obtained through single pulse transcranial magnetic stimulation. Ten suprathreshold (130% of RMT) stimuli will be delivered on primary motor cortex (C3).
5. Spinal cord activity: the level of excitability of spinal cord will be measured through the following outcomes:

   * Hoffman reflex (H reflex): the H reflex will be elicited by a percutaneous electrical stimulation on tibial nerve delivered on popliteal fossae and recorded the electromyographic responses from the soleus muscle. The values of maximal H reflex, M wave and maximal H reflex and maximal M wave ratio (H/M ratio) will be obtained through a recruitment curve. The recruitment curve will start with a stimulus intensity delivered from 2 milliampere (mA) and increasing on steps of 1 mA until to M wave curve stabilization (no increasing of the M wave amplitude).
   * Homosynaptic depression (HD): the HD will be obtained through a serie of two consecutive stimuli separated by a interstimulus interval (from 30ms until 10.000ms). The stimuli will be delivered on popliteal fossa and the electromyographic responses from soleus muscle will be recorded. The stimuli will be delivered with the intensity necessary to produce the maximal H reflex (this information will be available in the recruitment curve as stated before). The difference between the first and the second stimuli for each interstimulus interval will give rise to the recovery curve.
   * Nociceptive component of Withdrawal reflex (RIIIr): The RIIIr wil be elicited by delivering percutaneous electrical stimulation on sural nerve (behind the right lateral malleolus) and recording responses from the ipsilateral brevis head of the biceps femoris muscle. For the reflex threshold (RT) record, the initial current intensity will be adjusted to 2 mA and increased on steps of 1 mA, until obtain a response of at least 20 µV, accompanied by pain report. Then, 5 stimulus (130% RT) will be applied to obtain the latency and area average. Besides, pain perception will be controlled through an analogue scale graded from 0 (without perception of pain) to 10 points (greater pain already felt).
6. tsDCS: transcutaneous spinal cord stimulation will be delivered through a direct current (DC) stimulator (NeuroConn Plus, Germany) using a pair of saline-soaked sponge electrodes (35cm²). The active electrode (anode or cathode) will be placed between the eleventh and the twelfth thoracic vertebra) and the reference electrode, over the right arm (deltoid muscle). Will be delivered a current intensity of 2.5 mA, fade in and fade out of 10 seconds, during 20 minutes. Sham tsDCS has been used in several studies to evaluate active tsDCS effects. Sham tsDCS will be applied using the same electrodes placement and parameter settings of anodal tsDCS however, stimulation will last only 30 seconds but the volunteers will continue with electrodes montage for 20 minutes.Thus, early sensations (eg. mild to moderate tingling or itch) on stimulation site will be experienced without inducing any modulatory effects. Moreover, after each tsDCS session, an adverse effects questionnaire will be applied.
7. rTMS: Initially, the higher cortical representation area (hotspot) of first right dorsal interosseous (FDI) muscle will be determined through a figure-eight coil connected to the magnetic stimulator (Rapid2, Magstim, UK) held manually and positioned over the scalp (C3 - 10/20 System) at an angle of 45 degrees from the midline pointed to the target muscle (FDI). Thereafter, RMT will be measure. rTMS protocols was based on previous studies. Low frequency protocol: 1 hertz (Hz), 90% RMT, 1500 stimuli (1 train). High frequency protocol: 20 Hz, 90% RMT, 45 trains, 40 stimuli per train, inter interval of 28 seconds, 1800 stimuli. Sham rTMS will be performed with low frequency protocol using two coils. The first one - connected to the stimulator - will be positioned on a coil support close to the volunteer but not visible. Therefore, characteristic stimulation noises will be audible. The second - disconnected to the stimulator - will be placed over left primary motor area. After each rTMS session, presence of adverse effects will be computed.
8. Gait training: It consists of moderate gait training exercise for 20 minutes. To ensure that the exercise will be performed at moderate intensity will be used the 64% - 76% of maximum heart rate (HRmax = 220-age). Heart rate will be monitored every three minutes through a heart polar. In addition will be monitored perceived effort, gait speed and incline of the treadmill. The Borg scale will be used to evaluate perceived effort. This is an analogue scale graded from 6 (light exercise) to 20 points (exhaustive exercise). Information about the exercise on the treadmill will be noted in the evolution record.
9. Spinal cord activity: this evaluation will be performed immediately after (T0), thirty minutes after (T1) and 1 hour after (T2) the gait training. The procedures will be conducted following the same protocol.
10. Cortical brain activity: this evaluation will be performed after each revaluation of spinal cord activity (T0, T1 and T2). The procedures will be conducted following the same protocol.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed (assessed by Edinburgh Handedness Inventory)
* Healthy volunteers (self report)
* Sedentary or irregularly active (short version of the International Physical Activity Questionnaire)
* Contraceptive medication for women
* Without using drugs or neuroactive substances regularly

Exclusion Criteria:

* Pregnancy
* Presence of metallic implant close to the target stimulation area
* Acute eczema under the target stimulation area
* Pacemaker
* History of seizures or epilepsy
* Hemodynamic instability

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Changes on spinal excitability | six weeks (during stimulation protocol)
  Spinal excitability measures will be assessed by electrical stimulation of the tibial nerve (H-reflex and homosynaptic depression) and sural nerve (withdrawal reflex). The volunteer should stay in prone position for the stimulation of the tibial nerve (in the region of the popliteal fossa) and then in the lateral position for the stimulation of the sural nerve (in retromalleolar region).

SECONDARY OUTCOMES:
Changes on cortical brain activity (Intracortical inhibition) | six weeks (during stimulation protocol)
  The short intracortical inhibition (SICI) will be evaluated through pp-TMS. Subthreshold conditioning stimuli (80% of rest motor threshold - RMT) and suprathreshold test stimuli (130% of RMT) will be delivered at 3 milliseconds of interstimulus intervals (ISI). Ten stimuli will be applied at each condition (unconditioned pulse and pairs of stimuli with ISI of 3 milliseconds). Stimuli order delivery will be pseudo-randomized and SICI will be expressed as conditioned stimulus percentage regarding an unconditioned stimulus.
Changes on cortical brain activity (Intracortical facilitation) | six weeks (during stimulation protocol)
  The intracortical facilitation (ICF) will be evaluated through pp-TMS. Subthreshold conditioning stimuli (80% of RMT) and suprathreshold test stimuli (130% of RMT) will be delivered at 20 milliseconds of interstimulus intervals (ISI). Ten stimuli will be applied at each condition (unconditioned pulse and pairs of stimuli with ISI of 20 milliseconds). Stimuli order delivery will be pseudo-randomized and ICF will be expressed as conditioned stimulus percentage regarding an unconditioned stimulus.
Changes on cortical brain activity motor evoked potential (MEP) | six weeks (during stimulation protocol)
  The motor evoked potential (MEP) will be provided by ten unconditioned stimuli (130% RMT).

OTHER OUTCOMES:
Perceived of effort level | six weeks (during stimulation protocol)
  The Borg scale will be used to evaluate this measure. The volunteers will be enquired about their perceived of effort before, during (every three minutes) and after the gait training. Borg scale is an analogue scale graded from 6 (light exercise) to 20 points (exhaustive exercise).
Heart rate | six weeks (during stimulation protocol)
  To ensure that the exercise will be performed in a moderate intensity, the heart rate it will be monitored before, during (every three minutes ) and after the gait training by a cardiac polar.
Subjective perception of pain | six weeks (during stimulation protocol)
  the visual analog scale (VAS) will be apply to document the perception of pain. The VAS scores ranges from 0 (no perception of pain) to 10 (most pain I've felt).

CONTACTS AND LOCATIONS:
Overall Officials: Kátia K Monte-Silva, PhD, Study Director — Universidade Federal de Pernambuco
Locations (1):
- Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil